CLINICAL TRIAL: NCT04792437
Title: Research on Precise Immune Prevention and Treatment of Glioma Based on Multi-omics Sequencing Data
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yu Yao, MD (Other)
Responsible Party: Sponsor-Investigator, Yu Yao, MD, Professor, Huashan Hospital
Organization: Huashan Hospital (Other)
Other Study IDs: KY2021-059
Record Dates: First submitted 2021-03-01; First posted 2021-03-11 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Transcriptomics; Radiomics; Glioma
MeSH Terms: conditions — Glioma | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Peripheral blood、urine、feces、Glioma tissue、brain tissue、meninges、Cerebrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- glioma patients: glioma patients with routine surgery
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery — surgery

SUMMARY:
This project intends to use multiple types of biological samples from glioma patients and mouse intracranial tumor models as research objects, and comprehensively apply a series of omics sequencing technologies and molecular biology technologies to jointly define the following research objectives :

DETAILED DESCRIPTION:
1. Through high-throughput sequencing technologies such as， genome sequencing, transcriptome sequencing and single-cell sequencing, Proteomics，Metabonomics and Metagenomics， the similarities and differences of the glioma immune microenvironment within and between individuals were revealed from the multi-dimensional and big data level, and the immune molecular typing of glioma was established.
2. Establish and verify that the neoantigen polypeptides predicted by AI algorithm after analyzing multi-omics data (genome, transcriptome, etc.) have good killing effect on individual tumor cells.
3. To establish an intelligent evaluation model of glioma immunotyping by integrating imaging, pathology, high-throughput sequencing data and other omics information, and to provide a visual tool for monitoring changes in the intratumoral microenvironment of glioma patients, with the expectation of helping timely intervention of immunotherapy in patients with recurrence.

ELIGIBILITY:
Inclusion Criteria:

* The patients with glioma in the Department of Neurosurgery of Huashan Hospital Affiliated to Fudan University who meet the following three conditions can be enrolled

  1. They were 18-80 years old, male and female;
  2. The pathological diagnosis was glioma;
  3. On the basis of not affecting the clinical routine diagnosis, tissue (6 mm * 6 mm) or paraffin section (5 pieces) can be used for research;
  4. Sign informed consent or ethics committee approval

     Exclusion Criteria:

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing glioma surgery at Huashan Hospital
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival（OS），month | 24 month
  Survival time from surgery to death in 120 patients with glioma.
Progress Free Survival （PFS），month | 24 month
  Survival time from surgery to first progression or death from any cause in patients with glioma.
Tumor Mutation Burden（TMB），mutations/mb, drived from Genomic sequencing | 24 month
  the level of gene mutation，including TERT、GMEM、IDH.etc.
Reads Per Kilobase Million（RPKM），KB^(-1), drived from Transcriptome sequencing | 24 month
  the expression level of RNA,including mRNA、 miRNA、circRNA.etc
expression level of protein , drived from Protein sequencing | 24 month
  the expression level of protein, post-translational modification and protein-protein interaction，including PD1、PDL1、CD4、CD8.etc.
expression level of low molecular weight protein，drived from Metabonomics | 24 month
  the expression level and interaction of different Metabolites，including D-2-Hydroxyglutarate. etc.
expression level of DNA，drived from Metagenomics | 24 month
  Differences about DNA expression of all microorganisms in the environment
frequency of TCR/BCR clone，drived from Immunomics | 24month
  different expression level and interaction of Immune molecules，including TCR、BCR、antibody.etc.
expression level of protein，drived from paraffin-embedded specimens， retrospectively collected. | 24month
  different expression level of proteins in Gliomas with different grades and molecular subgroups (1000 cases)

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan hospital， Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ostrom QT, Gittleman H, Truitt G, Boscia A, Kruchko C, Barnholtz-Sloan JS. CBTRUS Statistical Report: Primary Brain and Other Central Nervous System Tumors Diagnosed in the United States in 2011-2015. Neuro Oncol. 2018 Oct 1;20(suppl_4):iv1-iv86. doi: 10.1093/neuonc/noy131. No abstract available. PMID 30445539
- [Background] Stupp R, Hegi ME, Mason WP, van den Bent MJ, Taphoorn MJ, Janzer RC, Ludwin SK, Allgeier A, Fisher B, Belanger K, Hau P, Brandes AA, Gijtenbeek J, Marosi C, Vecht CJ, Mokhtari K, Wesseling P, Villa S, Eisenhauer E, Gorlia T, Weller M, Lacombe D, Cairncross JG, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumour and Radiation Oncology Groups; National Cancer Institute of Canada Clinical Trials Group. Effects of radiotherapy with concomitant and adjuvant temozolomide versus radiotherapy alone on survival in glioblastoma in a randomised phase III study: 5-year analysis of the EORTC-NCIC trial. Lancet Oncol. 2009 May;10(5):459-66. doi: 10.1016/S1470-2045(09)70025-7. Epub 2009 Mar 9. PMID 19269895
- [Background] Tan AC, Ashley DM, Lopez GY, Malinzak M, Friedman HS, Khasraw M. Management of glioblastoma: State of the art and future directions. CA Cancer J Clin. 2020 Jul;70(4):299-312. doi: 10.3322/caac.21613. Epub 2020 Jun 1. PMID 32478924
- [Background] Chheda ZS, Kohanbash G, Okada K, Jahan N, Sidney J, Pecoraro M, Yang X, Carrera DA, Downey KM, Shrivastav S, Liu S, Lin Y, Lagisetti C, Chuntova P, Watchmaker PB, Mueller S, Pollack IF, Rajalingam R, Carcaboso AM, Mann M, Sette A, Garcia KC, Hou Y, Okada H. Novel and shared neoantigen derived from histone 3 variant H3.3K27M mutation for glioma T cell therapy. J Exp Med. 2018 Jan 2;215(1):141-157. doi: 10.1084/jem.20171046. Epub 2017 Dec 4. PMID 29203539
- [Background] Nejo T, Matsushita H, Karasaki T, Nomura M, Saito K, Tanaka S, Takayanagi S, Hana T, Takahashi S, Kitagawa Y, Koike T, Kobayashi Y, Nagae G, Yamamoto S, Ueda H, Tatsuno K, Narita Y, Nagane M, Ueki K, Nishikawa R, Aburatani H, Mukasa A, Saito N, Kakimi K. Reduced Neoantigen Expression Revealed by Longitudinal Multiomics as a Possible Immune Evasion Mechanism in Glioma. Cancer Immunol Res. 2019 Jul;7(7):1148-1161. doi: 10.1158/2326-6066.CIR-18-0599. Epub 2019 May 14. PMID 31088845
- [Background] Keskin DB, Anandappa AJ, Sun J, Tirosh I, Mathewson ND, Li S, Oliveira G, Giobbie-Hurder A, Felt K, Gjini E, Shukla SA, Hu Z, Li L, Le PM, Allesoe RL, Richman AR, Kowalczyk MS, Abdelrahman S, Geduldig JE, Charbonneau S, Pelton K, Iorgulescu JB, Elagina L, Zhang W, Olive O, McCluskey C, Olsen LR, Stevens J, Lane WJ, Salazar AM, Daley H, Wen PY, Chiocca EA, Harden M, Lennon NJ, Gabriel S, Getz G, Lander ES, Regev A, Ritz J, Neuberg D, Rodig SJ, Ligon KL, Suva ML, Wucherpfennig KW, Hacohen N, Fritsch EF, Livak KJ, Ott PA, Wu CJ, Reardon DA. Neoantigen vaccine generates intratumoral T cell responses in phase Ib glioblastoma trial. Nature. 2019 Jan;565(7738):234-239. doi: 10.1038/s41586-018-0792-9. Epub 2018 Dec 19. PMID 30568305
- [Background] Hilf N, Kuttruff-Coqui S, Frenzel K, Bukur V, Stevanovic S, Gouttefangeas C, Platten M, Tabatabai G, Dutoit V, van der Burg SH, Thor Straten P, Martinez-Ricarte F, Ponsati B, Okada H, Lassen U, Admon A, Ottensmeier CH, Ulges A, Kreiter S, von Deimling A, Skardelly M, Migliorini D, Kroep JR, Idorn M, Rodon J, Piro J, Poulsen HS, Shraibman B, McCann K, Mendrzyk R, Lower M, Stieglbauer M, Britten CM, Capper D, Welters MJP, Sahuquillo J, Kiesel K, Derhovanessian E, Rusch E, Bunse L, Song C, Heesch S, Wagner C, Kemmer-Bruck A, Ludwig J, Castle JC, Schoor O, Tadmor AD, Green E, Fritsche J, Meyer M, Pawlowski N, Dorner S, Hoffgaard F, Rossler B, Maurer D, Weinschenk T, Reinhardt C, Huber C, Rammensee HG, Singh-Jasuja H, Sahin U, Dietrich PY, Wick W. Actively personalized vaccination trial for newly diagnosed glioblastoma. Nature. 2019 Jan;565(7738):240-245. doi: 10.1038/s41586-018-0810-y. Epub 2018 Dec 19. PMID 30568303
- [Background] Li Y, Liu X, Xu K, Qian Z, Wang K, Fan X, Li S, Wang Y, Jiang T. MRI features can predict EGFR expression in lower grade gliomas: A voxel-based radiomic analysis. Eur Radiol. 2018 Jan;28(1):356-362. doi: 10.1007/s00330-017-4964-z. Epub 2017 Jul 28. PMID 28755054
- [Background] Grossmann P, Gutman DA, Dunn WD Jr, Holder CA, Aerts HJ. Imaging-genomics reveals driving pathways of MRI derived volumetric tumor phenotype features in Glioblastoma. BMC Cancer. 2016 Aug 8;16:611. doi: 10.1186/s12885-016-2659-5. PMID 27502180